CLINICAL TRIAL: NCT01746745
Title: Disposition of [14C]-LY2940680 Following Oral Administration in Healthy Subjects
Brief Title: A Study of LY2940680 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14892; I4J-MC-HHBF (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-12-07; First posted 2012-12-11 (Estimated); Results first posted 2019-07-22 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [^14C]-LY2940680 (Experimental): Single 100 milligram (mg) dose of LY2940680 containing 100 microCuries of carbon-14-labeled LY2940680 ([^14C]-LY2940680)
  Interventions: Drug: [^14C]-LY2940680

INTERVENTIONS:
Drug: [^14C]-LY2940680 — Administered as solution by mouth

SUMMARY:
This is a single dose study of radiolabelled LY2940680 taken by mouth in healthy participants to study how the body absorbs and removes LY2940680 from the blood. This study is for research purposes only and is not intended to treat any medical condition.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy sterile males or surgically sterile females or postmenopausal females, as determined by medical history and laboratory assessments
* Have a body mass index (BMI) of 18.5 to 32.0 kilograms per square meter (kg/m^2), inclusive

Exclusion Criteria:

* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Have consumed herbal supplements, grapefruit juice, grapefruits, grapefruit containing products, Seville orange juice, Seville oranges, star fruit, or star fruit juice within 7 days prior to dosing or intend to consume during the study
* Have donated blood of more than 500 milliliters (mL) within the last month
* Have participated in a [^14C]-study within the last 6 months prior to admission for this study
* Exposure to significant radiation within 12 months prior to dose (for example, serial X-ray or computed tomography scans, barium meal, current employment in a job requiring radiation exposure monitoring)
* Have a pattern less than once per 2 days to expel feces from the bowel through the rectum or acute constipation within 3 weeks of the day prior to dose

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants completed study at 14 days postdose or earlier if ≥90% of administered radioactivity recovered or 24-hour (h) urine and fecal samples from 2 consecutive collections each had radioactivity levels <1.0% of total administered radioactivity in urine and feces combined.
Groups:
- [^14C]-LY2940680: Single 100-milligram (mg) LY2940680 dose containing 100 microCuries of carbon-14-labeled LY2940680 ([^14C]-LY2940680), administered as an oral solution.
Period: Overall Study
Arm/Group | [^14C]-LY2940680
Started | 6
Received Study Drug | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Enrolled participants who received study drug and had at least 1 safety assessment postdose.
Groups:
- [^14C]-LY2940680: Single 100-mg LY2940680 dose containing 100 microCuries of [^14C]-LY2940680, administered as an oral solution.
Arm/Group | [^14C]-LY2940680
Number analyzed (Participants) | 6
Age, Customized [Count of Participants; unit: Participants]
  44 to 59 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Fecal Excretion of LY2940680 Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered
Description: The percentage of the total radioactive dose administered that was excreted in feces = [(amount of radioactivity recovered in feces)/(radioactive dose administered)]*100.
Time Frame: Predose up to 14 days postdose. Samples collected at 24-h intervals.
Population: Enrolled participants who received study drug and had evaluable pharmacokinetic (PK) data.
Measure: Mean (Standard Deviation); unit: percentage of dose administered
Arm/Group | [^14C]-LY2940680
Number analyzed (Participants) | 6
percentage of dose administered | 82.7 (2.81)

2. Primary Outcome: Urinary Excretion of LY2940680 Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered
Description: The percentage of the total radioactive dose administered that was excreted in urine=[(amount of radioactivity recovered in urine)/(radioactive dose administered)]*100.
Time Frame: Predose up to 14 days postdose. Samples collected at 6-h intervals on Day 1 (0-6, 6-12, and 12-24 h postdose) and at 24-h intervals thereafter.
Population: Enrolled participants who received study drug and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: percentage of dose administered
Arm/Group | [^14C]-LY2940680
Number analyzed (Participants) | 6
percentage of dose administered | 14.6 (1.68)

3. Secondary Outcome: Plasma PK of LY2940680 and LSN3185556: Maximum Observed Concentration (Cmax)
Description: The Cmax of LY2940680 and its equipotent active metabolite in the free base form, LSN3185556, is reported.
Time Frame: Predose up to 14 days postdose. Samples collected at 0.5, 1, 2, 3, 4, 6, 8, 10, and 12 h postdose on Day 1 and every 24 h thereafter
Population: Enrolled participants who received study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | [^14C]-LY2940680
Number analyzed (Participants) | 6
nanograms per milliliter (ng/mL)
  Plasma LY2940680 | 831 (6)
  Plasma LSN3185556 | 1210 (25)

4. Secondary Outcome: PK of Radioactivity: Cmax
Time Frame: as for outcome 3
Population: Enrolled participants who received study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram equivalents per gram (ng Eq/g)
Arm/Group | [^14C]-LY2940680
Number analyzed (Participants) | 6
nanogram equivalents per gram (ng Eq/g)
  Plasma Total Radioactivity | 2380 (7)
  Whole Blood Total Radioactivity | 1520 (6)

5. Secondary Outcome: PK of LY2940680, LSN3185556, and Radioactivity: Time of Maximum Observed Concentration (Tmax)
Description: The Tmax of LY2940680, LSN3185556, and total radioactivity in plasma are reported, as well as the Tmax for total radioactivity in whole blood.
Time Frame: as for outcome 3
Population: Enrolled participants who received study drug and had evaluable PK data.
Measure: Median (Full Range); unit: h
Arm/Group | [^14C]-LY2940680
Number analyzed (Participants) | 6
h
  Plasma LY2940680 | 1.51 [1.00 to 3.00]
  Plasma LSN3185556 | 2.50 [2.00 to 4.02]
  Plasma Total Radioactivity | 2.00 [1.00 to 3.00]
  Whole Blood Total Radioactivity | 2.00 [1.00 to 3.00]

6. Secondary Outcome: Plasma PK of LY2940680 and LSN3185556: Area Under the Concentration-Time Curve From Time 0 to the Last Time Point With a Measurable Concentration [AUC(0 to Tlast)]
Time Frame: as for outcome 3
Population: Enrolled participants who received study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter (ng*h/mL)
Arm/Group | [^14C]-LY2940680
Number analyzed (Participants) | 6
nanograms*hour per milliliter (ng*h/mL)
  Plasma LY2940680 | 5680 (19)
  Plasma LSN3185556 | 20400 (32)

7. Secondary Outcome: PK of Radioactivity: AUC(0 to Tlast)
Description: AUC(0 to Tlast) of total radioactivity in plasma and whole blood are reported in nanograms*hour equivalents per gram (ng*h Eq/g).
Time Frame: as for outcome 3
Population: Enrolled participants who received study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h Eq/g
Arm/Group | [^14C]-LY2940680
Number analyzed (Participants) | 6
ng*h Eq/g
  Plasma Total Radioactivity | 64800 (16)
  Whole Blood Total Radioactivity | 38200 (18)

8. Secondary Outcome: Relative Abundance of LY2940680 and the Metabolites of LY2940680 in Plasma
Description: Relative abundance was expressed and calculated as the percentage of plasma sample radioactivity=[(radioactivity in peak)/(radioactivity in sample)]*100. Metabolites with a relative abundance ≤6% are not reported.
Time Frame: Day 1 up to 3 days postdose. Samples collected at 2, 3, 4, 6, and 8 h postdose on Day 1 and every 24 h thereafter.
Population: Enrolled participants who received study drug and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: percentage of sample radioactivity
Arm/Group | [^14C]-LY2940680
Number analyzed (Participants) | 6
percentage of sample radioactivity
  LY2940680 (parent) | 11.1 (2.54)
  Metabolite M75 (LSN3185556) | 52.0 (5.14)
  Metabolite M63 | 17.1 (1.71)

9. Secondary Outcome: Relative Abundance of LY2940680 and the Metabolites of LY2940680 in Urine
Description: Relative abundance was expressed and calculated as the percentage of administered dose excreted in urine=[(percentage of radioactivity in peak)/100]*(percentage of dose in sample). Metabolites with a relative abundance ≤1% are not reported.
Time Frame: Predose up to 4 days postdose. Samples collected at 6-h intervals on Day 1 (0-6, 6-12, and 12-24 h postdose) and at 24-h intervals thereafter.
Population: Enrolled participants who received study drug and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: percentage of administered dose excreted
Arm/Group | [^14C]-LY2940680
Number analyzed (Participants) | 6
percentage of administered dose excreted
  LY2940680 (parent) | 0.105 (0.0937)
  Metabolite M43 | 2.87 (0.816)
  Metabolite M63 | 1.82 (0.740)

10. Secondary Outcome: Relative Abundance of LY2940680, the Metabolites of LY2940680, and LSN3185556 in Feces
Description: Relative abundance was expressed and calculated as the percentage of the administered dose excreted in feces=[(percentage of radioactivity in peak)/100]*(percentage of dose in sample). Metabolites with a relative abundance ≤1% are not reported.
Time Frame: Predose up to 8 days postdose. Samples collected at 24-h intervals.
Population: Enrolled participants who received study drug and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: percentage of administered dose excreted
Arm/Group | [^14C]-LY2940680
Number analyzed (Participants) | 6
percentage of administered dose excreted
  LY2940680 (parent) | 0.431 (0.313)
  Metabolite M43 | 37.1 (1.65)
  Metabolite M49 | 3.04 (0.861)
  Metabolite M73 | 3.19 (1.43)
  LSN3185556 | 2.90 (1.09)

ADVERSE EVENTS:
Arm/Group | [^14C]-LY2940680
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 3/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | [^14C]-LY2940680 (N=6)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days